CLINICAL TRIAL: NCT00815373
Title: A Comparative Analysis of the Effects of Cosopt® Versus Xalacom® on Ocular Hemodynamics and Intraocular Pressure in Patients With Primary Open-angle Glaucoma
Brief Title: The Effects of Cosopt® Vs Xalacom® on Ocular Hemodynamics and Intraocular Pressure (IOP) in Primary Open-angle Glaucoma (POAG)
Acronym: Xal-Cos
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants recruded.
Sponsor: Meir Medical Center (Other)
Responsible Party: Adi Abulafia, MD, Meir Medical Center, Kfar Saba, Affiliated to Tel Aviv University Israel
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 0155-08-MMC
Record Dates: First submitted 2008-12-09; First posted 2008-12-30 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Ocular Blood flow; Ocular hypertension; POAG; Ocular hemodynamics; Xalacom; Cosopt
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cosopt* b. i. d. (dosed morning and bedtime) will be administered topically
  Interventions: Drug: Dorzolamide+Timolol Maleate0.5%
- 2 (Active Comparator): Xalacom* q.d.(dosed bedtime) and placebo vehicle q.d. (dosed morning) topically in the other group
  Interventions: Drug: Latanoprost+Timolol Maleate0.5%+Lytears

INTERVENTIONS:
Drug: Dorzolamide+Timolol Maleate0.5% — Cosopt* b. i. d.
  Other Names: Cosopt
  Arms: 1
Drug: Latanoprost+Timolol Maleate0.5%+Lytears — Xalacom* QHS
  Other Names: Xalacom* QHS
  Arms: 2

SUMMARY:
Both Cosopt® and Xalatan® plus Timoptic® will significantly lower IOP, however only Cosopt® will demonstrate positive hemodynamic effects. The clinical significance of this will be investigated by examining the ophthalmic and short posterior ciliary arteries to determine the blood supply to the optic nerve head, the site of damage in glaucoma

DETAILED DESCRIPTION:
Background and Rationale

Apoptosis of retinal ganglion cell has been considered as the most plausible pathogenic mechanism of glaucoma. Apoptosis can be caused by neurotrophic factor withdrawal or glutamate release and both of them are triggered by elevated intraocular pressure (IOP) and ischemia simultaneously or separately.

The topical carbonic anhydrase inhibitor, Dorzolamide (Trusopt*), has recently been approved for chronic use in the treatment of glaucoma. The ocular hypotensive effects of this topical carbonic anhydrase inhibitor seem likely to produce the same results as *-adrenergic antagonists. Systemic carbonic anhydrase inhibitors are known to have vasodilatory effects (Maren,1987). Rassam S.M.B., Patel V. and Kohner E.M. (1993) have concluded that acetazolamide causes an increase in retinal blood flow in the human retinal circulation. It has also been demonstrated that Trusopt* increases retinal circulation as measured by scanning laser ophthalmoscopy (SLO) (Harris, Arend, Martin, 1996). Furthermore, Trusopt increases arteriovenous passage (AVP) time and improves contrast sensitivity in normal tension glaucoma patients (Harris, 1999).

Cosopt* (dorzolamide hydrochloride-timolol maleate ophthalmic solution) is combination of a topical carbonic anhydrase inhibitor and a topical beta-adrenergic receptor blocking agent. Each of these two components reduces intraocular pressure. The IOP-reducing effect of Cosopt b.i.d. was greater (1-3 mm Hg) than that of monotherapy with either 2.0 % dorzolamide t.i.d. or 0.5 % timolol b.i.d. The IOP-lowering effect of Cosopt* b.i.d. was approximately 1 mm Hg less than that of concomitant therapy with 2.0% dorzolamide t.i.d. and 0.5 % timolol b.i.d. A previous study showed that the retinal circulation (AVP time) was significantly accelerated after replacing Timoptic* with Cosopt* in glaucoma patients (Harris, 1999).

Latanoprost (Xalatan*) is a prostaglandin F2* analogue which is believed to reduce IOP by increasing the outflow of aqueous humor. The retinal vascular effects of Latanoprost, however, remain unclear. While some studies have shown PGF2* to induce constriction in bovine isolated aqueous veins (Nielsen 1996), other studies have been unable to demonstrate an effect on retrobulbar flow velocities (Drance 1996). It is possible that vasoconstrictive properties of the drug may produce a negative impact on previously ischemic retinal tissue or at best no change.

In a recent study comparing Trusopt® with Xalatan® some very encouraging results emerged, AVP time was significantly reduced with Trusopt®, but not with Xalatan® despite the fact that Xalatan® increases perfusion pressure (due to IOP) more than Trusopt®. This is the strongest evidence so far of a pressure independent effect of Trusopt® on ocular blood flow.

Objectives

* To compare the IOP efficacy of Cosopt® and Xalacom® on IOP.
* To determine the perfusion pressure effect of Cosopt® and Xalacom®.
* To determine the blood flow effect of the two drugs on the ophthalmic, central retinal and short posterior ciliary arteries, using Color Doppler Imaging (CDI).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater.
2. Patient signed an informed consent agreement.
3. Corrected visual acuity of 6/12 or better:
4. Characteristic glaucomatous visual-field loss and optic nerve head damage in one or both eyes.
5. Either IOP measurements ≥21 mmHg in the 3 months prior to study entry or IOP ≥ 21 mmHg at the end of the washout period
6. Patient on ≥1 IOP reducing agents. -

Exclusion Criteria:

1. Past history of ocular diseases (other than OAG / Cataract / Refractive error).
2. Past history of orbital/ocular surgery or trauma.
3. Receiving ≥ 3 IOP reducing agents.
4. Receiving agents known to produce significant cardiovascular, respiratory, renal or hepatic side effects.
5. Personal history of respiratory disease such as asthma, emphysema or other chronic obstructive pulmonary disease.
6. Personal history of congestive heart failure.
7. Personal history of bradycardia or 2nd and 3rd degree AV block.
8. Known allergy to sulfa.
9. Women who are pregnant or nursing.
10. Women who of child bearing age who are planning to become pregnant within one month after study completion.
11. Receiving Levitra, Viagra, Cialis or other erectile dysfunction drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Ocular hemodynamics as measured by Color Doppler imaging | 3 years

SECONDARY OUTCOMES:
Intraocular pressure as measured by Goldmann applanation tonometry | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Adi Abulafia, MD, Principal Investigator — Meir Medical Center, Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel